CLINICAL TRIAL: NCT02479126
Title: Interstitial Lung Diseases in the Veterans Administration Health System - A Retrospective Description of Patient Characteristics, Management, and Outcomes
Brief Title: Interstitial Lung Diseases in the Veterans Administration
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Robert Tighe (U.S. Federal Agency)
Collaborators: Durham VA Medical Center (U.S. Federal Agency); Boehringer Ingelheim (Industry)
Responsible Party: Sponsor-Investigator, Robert Tighe, Staff Physician, Durham VA Medical Center
Organization: Durham VA Medical Center (U.S. Federal Agency)
Other Study IDs: 01882
Record Dates: First submitted 2015-06-19; First posted 2015-06-24 (Estimated); Last update posted 2022-07-26 (Actual); Status verified 2022-07

CONDITIONS: Interstitial Lung Disease
Keywords: Interstitial Lung Disease; Idiopathic Pulmonary Fibrosis; Electronic Health Records; Computed Tomography; Mortality; Hospitalization; Acute care visits; Anti-inflammatory drug therapies
MeSH Terms: conditions — Lung Diseases, Interstitial; Idiopathic Pulmonary Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Interstitial Lung Disease: Patients will be identified from a specified 5 year period based on an International Classification of Diseases-9 (ICD-9) code diagnosis of Interstitial Lung disease (515) or Idiopathic Pulmonary Fibrosis (516.3). The patients will be obtained from the records of the Veterans Integrated Service Network (VISN) 6: VA Mid-Atlantic Health Care Network.

SUMMARY:
The primary objective of this research project is to describe the characteristics, diagnosis, management, and outcomes of patients with Interstitial Lung Disease (ILD) who received care at the Veteran's Administration Veterans Integrated Service Network (VISN) 6 Mid-Atlantic Health Care Network (VISN6) (includes North Carolina, Virginia and West Virginia) for up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Interstitial Lung Disease (ILD) ICD-9 code diagnosis 515.0 or 516.3

Exclusion Criteria:

* Inadequate documentation of patient receiving care for ILD in the health records

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adults with encounters at any VISN6 healthcare facility during specified time period
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2016-07; Primary Completion 2022-11 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Prevalence of Interstitial Lung Disease in the VISN6 Veterans Administration Patient Population | up to 5 years
Prevalence of Idiopathic Pulmonary Fibrosis in the VISN6 Veterans Administration Patient Population | up to 5 years

SECONDARY OUTCOMES:
Accuracy of ICD-9 Codes for diagnosis of Interstitial Lung Disease | up to 5 years
  Will compare the reported ICD-9 code diagnosis with the diagnosis made after chart review and re-interpretation of the lung imaging and pathology
Frequency of ICD-9 code diagnosis of Interstitial Lung Disease and clinic consultation with a pulmonary provider | up to 5 years
Prevalence of Co-morbid Diabetes Mellitus with Interstitial Lung Disease | up to five years
  Compare the prevalence of diabetes with interstitial lung disease as compared to the prevalence of diabetes in the general VA population

CONTACTS AND LOCATIONS:
Overall Officials: Robert M Tighe, MD, Principal Investigator — Duke University Department of Medicine and Durham VA Medical Center
Locations (1):
- Durham VA Medical Center, Durham, North Carolina, United States